CLINICAL TRIAL: NCT03450733
Title: Post-Market Surveillance of the Wright Medical Technology Metal-on-Metal Total Hip System (FDA 522 Order)
Brief Title: Wright Medical Technology Metal-on-Metal 522 Post-Market Surveillance Study
Status: Completed | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11LJH001
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Hip; Hip Disease; Hip Osteoarthritis; Joint Pain
Keywords: Metal-on-Metal; MOM; Total Hip Arthroplasty; THA
MeSH Terms: conditions — Osteoarthritis, Hip; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood and serum samples will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Previously Implanted (Group 1): Subjects previously implanted with components of the Wright Medical Technology (WMT) Metal-on-Metal (MoM) Total Hip Arthroplasty (THA) System
  Interventions: Device: Wright Medical Technology Metal-on-Metal Total Hip System
- Control (Group 2): Control, non-implanted subjects

INTERVENTIONS:
Device: Wright Medical Technology Metal-on-Metal Total Hip System — Subjects in Group 1 previously implanted prior to the study start date will be identified from Investigator records. Collected data will be evaluated in aggregate and cross-sectioned by year of implantation. Subjects will be cross-sectioned by the time that has elapsed between implantation and the initial visit (e.g. 5 years, 6 years) using contiguous visit windows (number of years + 6 months). Subject data will be grouped in order to create cross-sectional epochs of ≤ 8 years and > 8 years.
  Groups: Previously Implanted (Group 1)

SUMMARY:
This study is in response to the Food and Drug Administration (FDA) call to all manufacturers with 510(k) clearance for metal-on-metal (MoM) total hip arthroplasty (THA) devices to conduct postmarket surveillance studies. MicroPort has various acetabular shells, acetabular liners, fixation screws, femoral heads, femoral stems, modular necks, and proximal bodies currently cleared for MoM indications. Together these components comprise the Wright Medical Technology (WMT) MoM THA System. The primary objective of the study is to determine the incidence of adverse local tissue reactions (ALTR) in each THA implanted with the WMT MoM THA System overall and to create cross-sectional epochs of ≤ 8 years and > 8 years, since implantation.

ELIGIBILITY:
Inclusion Criteria:

To be included in Group 1, subjects must meet all of the following criteria:

1. Has been implanted with appropriate components of the WMT MOM THA System
2. Has previously undergone primary THA for any of the following:

   1. non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, or avascular necrosis;
   2. inflammatory degenerative joint disease including rheumatoid arthritis;
   3. correction of functional deformity.
3. Is willing and able to complete required study visit(s) and assessments
4. Plans to be available for the required study visit
5. Is capable of providing sufficient blood for sampling according to blood draw procedures
6. Is willing to sign the approved Informed Consent document

Previously implanted bilateral subjects can have both THAs enrolled in the study provided: 1) the specified combination of components were implanted in both, 2) all other aspects of the Inclusion/Exclusion Criteria are satisfied, 3) enrollment does not exceed the subject count specified in the Clinical Trial Agreement and protocol enrollment strategy, and 4) the subject agrees to a second Informed Consent document and data collection specific to the second THA. Enrollment and treatment of a previously unimplanted hip is not permitted in this study.

To be included in Group 2, subjects must meet all of the following criteria:

1. Does not have a metal implant (total hip, total knee, spinal, etc.) with the exception of dental implants
2. Is not an employee of the Investigator
3. Is willing and able to provide Informed Consent document
4. Is willing and able to attend the requested study visit(s) and assessments
5. Is capable of providing sufficient blood for sampling according to blood draw procedures

Exclusion Criteria:

Subjects will be excluded from either study group if they meet any of the following criteria:

1. Subject is currently enrolled in another clinical investigation which could affect the endpoints of this protocol
2. Subject is unwilling or unable to sign the Informed Consent document
3. Subject has documented substance abuse issues
4. Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
5. Subject is currently incarcerated or has impending incarceration
6. Group 1 only: Subject has a condition or previously implanted medical device that contraindicates MRI (e.g. pacemaker, implantable defibrillator)
7. Group 1 only: Subject was skeletally immature (less than 21 years of age) at time of implantation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Subjects previously implanted with components of the Wright Medical Technology (WMT) Metal-on-Metal (MoM) Total Hip Arthroplasty (THA) System
  Group 2: Control, non-implanted subjects
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Local Tissue Reactions (ALTR) | ≤ 8 years and > 8 years, since implantation
  To determine the incidence rate of ALTR in subjects implanted with WMT MoM THA System (Group 1)

SECONDARY OUTCOMES:
Determine chromium and cobalt whole blood and serum ion levels across time intervals | ≤ 8 years and > 8 years, since implantation
  Cobalt and chromium metal ion levels will be measured in whole blood and serum from subjects implanted with the WMT MoM THA System (Group 1) at each defined cross-section interval.
Establish baseline for chromium and cobalt whole blood and serum ion levels across time intervals | ≤ 8 years and > 8 years, since implantation
  Analyze difference in chromium and cobalt whole blood and serum ion levels in subjects implanted with the WMT MoM THA System (Group 1) versus control subjects (Group 2) cross-sectionally.
Compare functional outcomes of subjects implanted with the WMT MoM THA System with and without ALTR (Group-1 subjects). | ≤ 8 years and > 8 years, since implantation
  Calculate and compare composite hip outcomes scores, via the validated HOOS scores, in Group 1 subjects with ALTR versus Group 1 subjects without ALTR
Compare cobalt and chromium metal ion levels in subjects implanted with the WMT MoM THA System with and without ALTR (Group-1 subjects). | ≤ 8 years and > 8 years, since implantation
  Analyze difference in cobalt and chromium metal ion levels from Group 1 subjects with ALTR versus Group 1 subjects without ALTR

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - TriWest Research Associates, El Cajon, California
  - BioSolutions Research Center, La Mesa, California
  - University of Iowa, Iowa City, Iowa
  - Spokane Joint Replacement Center, Inc., Spokane, Washington